CLINICAL TRIAL: NCT00408928
Title: Phase II Trial of VELCADE® (Bortezomib) for Steroid Refractory Acute GVHD
Brief Title: Study on the Safety and Effectiveness of VELCADE® in the Treatment of Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04U.177; 2004-19 (Other: CCRRC); JT 1129 (Other: JeffTrial Number)
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Graft-versus-Host Disease
Keywords: Graft-versus-Host Disease; bortezomib
MeSH Terms: conditions — Graft vs Host Disease | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib for Treatment of GHVD (Experimental): To determine if bortezomib (VELCADE®) will successfully inhibit T-cell responses in clinically acute graft-versus-host disease (GVHD) after allogeneic hematopoietic stem cell transplantation (HSCT).
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib at 1.3 mg/m2/dose given twice weekly for two weeks followed by a 10-day rest period. If patients have a complete response, they will receive additional cycles of bortezomib.
  Other Names: VELCADE; PS-341

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of VELCADE® in the treatment of acute graft-versus-host disease (GVHD) that has not responded to steroids or has worsened when the steroid dose was decreased. VELCADE® is a drug that inhibits certain immune reactions that happen when lymphocytes encounter foreign substances. We are doing this research to determine if VELCADE® may be useful in treating GVHD.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) is a serious complication after bone marrow transplantation from another donor. GVHD is caused by certain cells called lymphocytes. Normally these cells make immune reactions that help protect the body from foreign substances that cause infection. Here, these cells attack the normal tissues of the body as if they were foreign substances. This interferes with the normal function of vital organs and results in their damage. In GVHD these cells attack the skin, liver and bowel. GVHD also increases the chances of infection.

VELCADE® is a drug that inhibits certain immune reactions that happen when lymphocytes encounter foreign substances. We are doing this research to determine if VELCADE® may be useful in treating GVHD.

VELCADE® is approved by the Food and Drug Administration (FDA) for the treatment of multiple myeloma in patients who have received at least two prior therapies and have demonstrated disease progression on their last therapy. Its effectiveness is also being tested in other cancers. The dose of the drug being used in this research study is the same as what is used for the treatment of multiple myeloma. It has not been approved by the FDA for use in GVHD. Therefore, using VELCADE® for GVHD is experimental in this research study.

ELIGIBILITY:
Inclusion Criteria: (All criteria must be met)

1. Patients must have undergone an allogeneic HSCT
2. Clinical or histological evidence of AGVHD
3. Has been treated with a minimum of 2mg/kg of methylprednisolone per day or equivalent dose of steroids and either one of the following:

   1. Has had a minimum of 3 days of steroids including the day of assignment and has progressive disease.
   2. Has had a minimum of 7 days of steroids including the day of assignment and has had no response.
   3. AGVHD progresses at anytime when steroids are tapered to less than 2mg/kg/day of methylprednisolone or its equivalent.
4. Performance status ECOG 0-2
5. Patients must be willing to use contraception if they have childbearing potential
6. Able to give informed consent
7. Patients must be > 18 years of age, with no upper age limit.

Exclusion Criteria: (Any one criteria will exclude patient)

1. Performance status of ECOG >2.
2. >Grade3 peripheral neuropathy at the time of enrollment
3. Patient has a creatinine clearance (calculated or measured) of <30mL/min at the time of enrollment.
4. Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry , any ECG abnormality at Screening has to be documented by the investigator/co-investigator as not medically relevant.
5. Patient has hypersensitivity to bortezomib, boron or mannitol.
6. Female subject is pregnant or breast-feeding.
7. Patient has received other investigational drug within 14 days prior to enrollment.
8. Serious medical or psychiatric illness likely to interfere with participation in this clinical study or to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Wagner, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospital — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib for Treatment of GHVD: Bortezomib at 1.3 mg/m2/dose given twice weekly for two weeks followed by a 10-day rest period. If patients have a complete response, they will receive additional cycles of bortezomib.
Period: Overall Study
Arm/Group | Bortezomib for Treatment of GHVD
Started | 11
Completed | 8
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Infection indistinguishable from GVHD | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib for Treatment of GHVD
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.68 (15.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Response to Bortezomib (VELCADE®)
Description: Response is the primary endpoint of this study and will be scored on day 21 (3 weeks after the first dose of VELCADE) and every 3 weeks subsequently. Patients who progress or expire before the end of the study will be considered non-responders.
  Patients are evaluated for response in an organ if they have AGVHD in that organ at the start of treatment with VELCADE or if AGVHD develops after the start of VELCADE, but before the time period of evaluation. Complete response in an organ is defined as no evidence clinical or biochemical signs of AGVHD. For the overall assessment, it is defined as complete resolution of rash, abnormal LFTs, and absence of diarrhea attributed to AGVHD.
  Partial response is defined as a one stage decrease in any organ system without worsening in other organ systems.
Time Frame: Through 30 days post-treatment
Measure: Number; unit: participants
Arm/Group | Bortezomib for Treatment of GHVD
Number analyzed (Participants) | 8
participants
  Complete response | 2
  Partial response | 2
  No response | 4

2. Secondary Outcome: Number of Toxicities Related to Bortezomib (VELCADE®)
Description: Observe the toxicities of VELCADE® when administered to recipients of allogeneic hematopoietic stem cell transplant in the setting of steroid refractory or steroid dependent acute graft-versus-host disease.
Time Frame: Through 30 days post-traeatment
Measure: Number; unit: toxicities
Arm/Group | Bortezomib for Treatment of GHVD
Number analyzed (Participants) | 8
toxicities | 18

ADVERSE EVENTS:
Arm/Group | Bortezomib for Treatment of GHVD
Serious Adverse Events (participants affected / at risk) | 9/11
Other Adverse Events (participants affected / at risk) | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib for Treatment of GHVD (N=11)
Nausea (General disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Diarrhea (General disorders) | 4 (5)
GVHD (General disorders) | 1 (1)
Hypotension (General disorders) | 1 (1)
Seizure (General disorders) | 1 (1)
Cystitis (General disorders) | 1 (1)
Lack of appetite (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 1 (1)
Infection (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib for Treatment of GHVD (N=11)
Neuropathy (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes